CLINICAL TRIAL: NCT05488353
Title: A Clinical Study of Disitamab Vedotin for Injection Combined With Penpulimab Injection in Neoadjuvant Therapy for Patients With HER2-expressing Cisplatin-intolerant cT2-T4aNxM0 Bladder Urothelial Carcinoma
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other); Nanfang Hospital, Southern Medical University (Other); Southern Medical University, China (Other); The Third Affiliated Hospital of Southern Medical University (Other Government)
Responsible Party: Principal Investigator, Lin Tianxin, chief physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C039
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Bladder Cancer
Keywords: HER2-expressing; Cisplatin-intolerant; Disitamab Vedotin for Injection; Penpulimab Injection
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — disitamab vedotin; Injections; penpulimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Disitamab Vedotin for Injection, 2.0 mg/kg, given as an IV infusion on day 1, and Penpulimab Injection, 200 mg, on every 21 days On day 1 of the cycle, it is given as an intravenous infusion. Order of use: Disitamab Vedotin for Injection → Penpulimab Injection.
  Interventions: Drug: Disitamab Vedotin for Injection,Penpulimab Injection

INTERVENTIONS:
Drug: Disitamab Vedotin for Injection,Penpulimab Injection — After completion of all screening activities, patients confirmed to be eligible will enter the study and receive the following treatments.
  Neoadjuvant regimen (up to 4 cycles): Disitamab Vedotin for Injection, 2.0 mg/kg, given as an IV infusion on day 1, and Penpulimab Injection, 200 mg, on every 21 days On day 1 of the cycle, it is given as an intravenous infusion. Order of use: Disitamab Vedotin for Injection → Penpulimab Injection.

SUMMARY:
This study is a one-arm exploratory clinical study of Disitamab Vedotin for Injection combined with Penpulimab Injection designed for cisplatin intolerant CT2-T4anxm0 bladder urothelial carcinoma patients.It will confirme the efficacy and safety of Disitamab Vedotin for Injection combined with Penpulimab Injection neoadjuvant treatment for cisplatin intolerant CT2-T4anxm0 bladder urothelial carcinoma patients. Finally, it will provide new evidence-based medical evidence for neoadjuvant therapy for such patients.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, single-arm prospective clinical study to evaluate the neoadjuvant treatment of Disitamab Vedotin for Injection combined with Penpulimab Injection in cisplatin-intolerant cT2-T4aNxM0 bladder urothelial carcinoma Efficacy and safety in patients. If the subject does not withdraw from the trial voluntarily, the toxic and side effects caused by the drug are intolerable, or the investigator believes that the subject is not suitable for further trials, each subject will undergo the following treatment after surgery, and in Efficacy evaluation and follow-up were performed in each cycle.

After completion of all screening activities, patients who are identified as eligible will enter the study and receive the following treatments and visits: Neoadjuvant therapy with Disitamab Vedotin for Injection combined with Penpulimab Injection (administered for a maximum of 4 cycles), every three One week is a medication cycle; patients received radical cystectomy after neoadjuvant chemotherapy; postoperative pathological complete remission rate, downstaging rate, and regular follow-up for two years were evaluated to evaluate the safety of the patients drugs/surgery, and to evaluate the patients new Survival after curative resection with adjuvant immunotherapy combined with chemotherapy.

Neoadjuvant regimen (up to 4 cycles): Disitamab Vedotin for Injection, 2.0 mg/kg, given as an IV infusion on day 1, and Penpulimab Injection, 200 mg, on every 21 days On day 1 of the cycle, it is given as an intravenous infusion. Order of use: Disitamab Vedotin for Injection → Penpulimab Injection.

Surgical plan: radical cystectomy + urinary diversion.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this trial, be able to sign a written informed consent form, and understand and agree to comply with the requirements of this study and the evaluation schedule.
2. The age on the date of signing the informed consent form is 18 to 75 years old.
3. If it is a patient with cT2-T4aNxM0 bladder urothelial carcinoma with histological diagnosis and imaging evaluation based on AJCC eighth edition bladder cancer TNM staging, if the investigator believes that there is residual disease after TURBT surgery; the histology is mixed type. Oncological patients require urothelial carcinoma predominance (at least 50%).
4. Patients who are intolerant or not receiving cisplatin must be determined by the investigator. Patients who do not tolerate cisplatin chemotherapy must meet at least one of the following criteria:

   1. The performance status of ECOG is >1;
   2. Creatinine clearance rate < 60mL/min;
   3. Hearing loss ≥ grade 2 in the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) 5th edition;
   4. Peripheral neuropathy grade ≥ 2 in NCI-CTCAE 5th edition;
   5. Suffering from New York Heart Association grade 3 or higher heart failure.
5. According to the assessment by the investigator, the need for radical cystectomy after neoadjuvant therapy, and the indications for radical cystectomy are met, and they are willing to undergo the surgery.
6. HER2 testing at local laboratory using pre-treatment tumor specimens: HER2 expression confirmed after IHC results (defined as: IHC 1+ 2+ 3+).
7. ECOG fitness status 0~1.
8. The patient's organ function is good, as measured by the following screening laboratory values ??(obtained ≤14 days prior to enrollment):

   a. Patients should not be on growth factor support ≤ 14 days prior to sample collection when screening for: i. Absolute neutrophil count ≥1.5×109/L; ii. Platelets≥100×109/L; iii. Hemoglobin≥90g/L; b. International normalized ratio or activated partial thromboplastin time ≤ 1.5 upper limit of normal (ULN); c. Serum total bilirubin≤1.5×ULN; d. AST, ALT and alkaline phosphatase≤2.5×ULN; e. The calculated creatinine clearance rate is greater than 30 mL/min;
9. Non-conceptual or fertile women must be willing to use highly effective contraception during the study period and for ≥ 120 days after the last dose of Vidicitumumab or Piamprizumab (whichever occurs later), and Negative urine or serum pregnancy test results within ≤7 days prior to enrollment.
10. Non-sterilized males must be willing to use highly effective contraception during the study period and for ≥ 120 days after the last dose of vildicotumab or pianiprilumab (whichever occurs later).

Exclusion Criteria:

1. Previously received therapies targeting PD-1, PD-L1, PD-L2, CTLA4, Her2 or other antibodies or drugs that specifically target T cell co-stimulation or checkpoint channels.
2. Received other approved systemic anticancer therapy or systemic immunomodulators (including but not limited to interferon, interleukin 2 and tumor necrosis factor) within 28 days before enrollment.
3. Previously received radiotherapy for bladder cancer.
4. Received drug treatment for tumors in the past, except for the following:

   1. For patients who have received systemic chemotherapy in the past, a treatment-free interval of at least 12 months from the last treatment to the start of neoadjuvant drug therapy;
   2. Local intravesical chemotherapy or immunotherapy ended at least 1 week before the initiation of study neoadjuvant drug therapy.
5. Major surgery or major trauma within 28 days before enrollment (implantation of vascular access device and TURBT are not considered major surgery).
6. Serious infection requiring systemic antibacterial, antifungal or antiviral treatment within 14 days before enrollment (HBV infection is performed according to the instructions of exclusion criterion 12).
7. Have been vaccinated with live vaccines within 28 days before enrollment (seasonal influenza vaccines are usually inactivated vaccines, so they are allowed to be used. Intranasal vaccines are live vaccines, so they are not allowed to be used).
8. Received any Chinese herbal medicine or proprietary Chinese medicine for cancer control within 14 days before enrollment.
9. Active autoimmune disease that requires systemic treatment, and the investigator evaluates that it has an impact on the study treatment.
10. Long-term use of large amounts of hormones or other immunosuppressive agents is required, and the investigator evaluates that it has an impact on the study treatment.
11. History of potassium, sodium, calcium abnormalities or hypoalbuminemia, interstitial lung disease, non-infectious pneumonia, or other uncontrolled systemic diseases, including diabetes, hypertension, cardiovascular disease, that the investigator believes may affect treatment (such as active heart disease within 6 months before enrollment, including: severe/unstable angina pectoris, myocardial infarction, symptomatic congestive heart failure and ventricular arrhythmia requiring drug treatment, etc.), etc.
12. Untreated chronic hepatitis B subjects or hepatitis B virus (HBV) carriers with HBV DNA ≥ 500 IU/mL (2500 copies/mL) are not allowed to enter the study. Note: Inactive hepatitis B surface antigen carriers or patients with stable active HBV infection (HBV DNA <500 IU/mL [2500 copies/mL]) after continuous antiviral therapy can be enrolled. HBV DNA testing is performed only in patients who are positive for antibodies to hepatitis B surface antigen.
13. Patients with active hepatitis C are not eligible. Patients who tested negative for HCV antibodies during the screening period, or those who tested negative for HCV RNA after positive HCV antibody tests could be enrolled. Only patients who test positive for HCV antibodies require HCV RNA testing.
14. A history of immunodeficiency (including positive human immunodeficiency virus HIV test, other acquired and congenital immunodeficiency diseases) or a history of allogeneic stem cell transplantation or organ transplantation.
15. Known hypersensitivity to other monoclonal antibodies.
16. Known allergy to any study drug or excipient.
17. Concurrently participate in another therapeutic clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 12 months
  As assessed by the investigator,proportion of patients without residual tumor lesion among patients who underwent radical cystectomy after completion of clinical trial treatment.

SECONDARY OUTCOMES:
pathological downstaging rate | 12 months
  The pathological downstaging rate is judged according to the pathological results after surgery whether the downstaging is below T2 stage.
safety evaluation | up to 3 years
  Safety is evaluated by monitoring and recording all adverse events graded as NCI-CTCAE V5.0 or Clavien-Dindo.
EFS EFS | up to 3 years
  Event-free survival (EFS) is the time from the start of the first neoadjuvant therapy to disease progression, death from any cause, or new development of other tumors.
OS | up to 3 years
  Overall survival (OS) is defined as the time from the start of treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Tianxin Lin, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] preliminary safety and efficacy results of RC48 combined with toripalimab in patients wit local advaned or metastatic Urothelial carcinoma(NCT04264936,RC48-C014)
- [Background] An Open-label, Single-arm, Multicenter, Phase II Study of RC48 to Evaluate the Efficacy and Safety of Subjects With HER2 Overexpressing Locally Advanced or Metastatic Urothelial Cancer (NCT03809013,RC48-C009)
- [Background] Sheng X, Yan X, Wang L, Shi Y, Yao X, Luo H, Shi B, Liu J, He Z, Yu G, Ying J, Han W, Hu C, Ling Y, Chi Z, Cui C, Si L, Fang J, Zhou A, Guo J. Open-label, Multicenter, Phase II Study of RC48-ADC, a HER2-Targeting Antibody-Drug Conjugate, in Patients with Locally Advanced or Metastatic Urothelial Carcinoma. Clin Cancer Res. 2021 Jan 1;27(1):43-51. doi: 10.1158/1078-0432.CCR-20-2488. Epub 2020 Oct 27. PMID 33109737
- [Background] Antitumor activity of neoadjuvant treatment with enfortumab vedotin monotherapy in patients with muscle invasive bladder cancer (MIBC) who are cisplatin-ineligible

DOCUMENTS (2):
  • Study Protocol (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT05488353/Prot_000.pdf
  • Informed Consent Form (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT05488353/ICF_001.pdf